CLINICAL TRIAL: NCT02394340
Title: An Open-Label, Maximal Use Study Evaluating the Drug Interaction Potential of Luliconazole Cream 1% in Subjects With Tinea Pedis and Tinea Cruris
Brief Title: Study Evaluating the Drug Interaction Potential of Luliconazole Cream 1% in Participants With Tinea Pedis and Tinea Cruris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-1012
Record Dates: First submitted 2015-02-19; First posted 2015-03-20 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Tinea Pedis; Tinea Cruris
MeSH Terms: conditions — Tinea Pedis; Tinea Cruris | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Luliconazole Cream 1% (Experimental): Participants will receive 1 oral capsule of omeprazole 40 milligrams (mg) on Day 1 and Day 8. Participants will also receive luliconazole cream 1% to cover the entire affected surface areas and adjacent areas once daily in the morning on Day 2 (24 hours after initial omeprazole dosing) through Day 8.
  Interventions: Drug: Omeprazole 40 mg; Drug: Luliconazole Cream 1%

INTERVENTIONS:
Drug: Omeprazole 40 mg — Oral capsule to be taken as per the instructions regarding proper dosing technique.
Drug: Luliconazole Cream 1% — Topical cream to be applied as per the instructions regarding proper study drug application technique.
  Other Names: LUZU Cream 1%

SUMMARY:
This is an open-label, maximal use study to evaluate whether luliconazole in plasma acts as an inhibitor of cytochrome P2C19 (CYP2C19) as measured by circulating levels of omeprazole before and after treatment with a maximum dose of luliconazole cream 1% in participants with moderate to severe tinea pedis and tinea cruris.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a clinical diagnosis of moderate to severe interdigital tinea pedis, as defined by a Physician's Global Assessment (PGA) score of 2 or 3 on both feet, and moderate to severe tinea cruris, as defined by a PGA score of 2 or 3
* Participants with a mycological diagnosis of tinea pedis and tinea cruris confirmed by the detection of fungal hyphae on a microscopic potassium hydroxide (KOH) wet mount
* Participants must be in good general health and free of any disease that might interfere with study evaluations
* Participants with the ability and willingness to follow all study procedures, attend all scheduled visits, and successfully complete the study

Exclusion Criteria:

* Female participants who are pregnant and/or nursing or planning a pregnancy during the course of the trial
* Participants who are immunocompromised
* Participants who have a recent history of or currently known drug or alcohol abuse
* Participants with a history of intolerance or hypersensitivity to imidazole compounds, proton pump inhibitors, or the inactive components of luliconazole cream 1% or omeprazole
* Participants with a life-threatening condition within the last 6 months
* Participants with uncontrolled diabetes mellitus
* Participants who are unable to communicate or cooperate with the Investigator
* Participants using medications for treatment of tinea pedis and/or tinea cruris (see Investigator for length of time prior to study start)
* Participants receiving concomitant drugs that are known to inhibit and/or induce CYP2C19 and/or CYP3A4, or that interact with omeprazole
* Because of the potential for drug interaction with luliconazole, administration with medications that are known to be substrates of CYP3A4, CYP2B6, CYP2C8, and CYP2C19 should be carefully monitored

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Americas, Inc.
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Luliconazole Cream 1%: Participants received 1 oral capsule of omeprazole 40 milligrams (mg) on Day 1 and Day 8. Participants also received luliconazole cream 1% to cover the entire affected surface areas and adjacent areas once daily in the morning on Day 2 (24 hours after initial omeprazole dosing) through Day 8.
Period: Overall Study
Arm/Group | Luliconazole Cream 1%
Started | 20
Received at Least 1 Dose of Study Drug | 20
Completed | 18
Not Completed | 2
Not completed — Failed drug screen test | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 application of study drug and had at least 1 post-Baseline assessment.
Groups:
- Luliconazole Cream 1%: Participants received 1 oral capsule of omeprazole 40 mg on Day 1 and Day 8. Participants also received luliconazole cream 1% to cover the entire affected surface areas and adjacent areas once daily in the morning on Day 2 (24 hours after initial omeprazole dosing) through Day 8.
Arm/Group | Luliconazole Cream 1%
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.05 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Circulating Levels (Plasma Concentration) of Omeprazole Prior to Treatment With Luliconazole Cream 1%
Description: Circulating plasma levels of omeprazole were measured using validated liquid chromatography with tandem mass spectrometry detection (LS/MS-MS) methods. The range for omeprazole determination was 4.64-9.27 nanograms/milliliter (ng/mL). Serial blood sampling occurred in each enrolled participant up to 24 hours post treatment (Day 1) with omeprazole (before the start of luliconazole cream 1% treatment on Day 2).
Time Frame: 15 minutes predose; 15, 30, 45, and 60 minutes postdose; and 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 24 hours postdose of omeprazole on Day 1
Population: Randomized participants who received at least 1 dose of study drug and had evaluable data at the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Luliconazole Cream 1%
Number analyzed (Participants) | 20
ng/mL
  Predose | 0 (0)
  15 minutes postdose | 0 (0)
  30 minutes postdose | 23.67 (89.46)
  45 minutes postdose | 196.30 (301.31)
  1 hour postdose | 463.74 (546.51)
  1.5 hours postdose | 526.98 (499.60)
  2 hours postdose | 655.70 (520.31)
  2.5 hours postdose | 621.08 (464.55)
  3 hours postdose | 636.60 (508.53)
  4 hours postdose | 468.79 (355.49)
  6 hours postdose | 235.20 (214.29)
  8 hours postdose | 129.70 (129.08)
  10 hours postdose | 74.24 (84.54)
  24 hours postdose | 3.32 (6.18)

2. Primary Outcome: Circulating Levels (Plasma Concentration) of Omeprazole After 1 Week of Treatment With Luliconazole Cream 1%
Description: Circulating plasma levels of omeprazole were measured using validated LS/MS-MS methods. The range for omeprazole determination was 4.64-9.27 ng/mL. Serial blood sampling occurred in each enrolled participant up to 24 hours post treatment (Day 8) with omeprazole (after using luliconazole cream 1% treatment for 1 week).
Time Frame: 15 minutes predose; 15, 30, 45, and 60 minutes postdose; and 1.5, 2, 2.5, 3, 4, 6, 8, 10, and 24 hours postdose of omeprazole on Day 8
Population: Randomized participants who received at least 1 dose of study drug and had evaluable data at the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Luliconazole Cream 1%
Number analyzed (Participants) | 18
ng/mL
  Predose | 0 (0)
  15 minutes postdose | 0 (0)
  30 minutes postdose | 18.11 (68.24)
  45 minutes postdose | 142.72 (298.29)
  1 hour postdose | 317.21 (401.97)
  1.5 hours postdose | 637.56 (509.09)
  2 hours postdose | 763.51 (607.80)
  2.5 hours postdose | 700.91 (423.74)
  3 hours postdose | 730.56 (349.10)
  4 hours postdose | 586.83 (309.83)
  6 hours postdose | 323.40 (219.50)
  8 hours postdose | 190.15 (154.82)
  10 hours postdose | 111.51 (102.30)
  24 hours postdose | 6.84 (10.01)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 9
Description: All participants who received at least 1 application of study drug and had at least 1 post-Baseline assessment.
Arm/Group | Luliconazole Cream 1%
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luliconazole Cream 1% (N=20)
Muscle strain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate Aminotransferase increased (Investigations) | 1
Hemoglobin decreased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study was designed to test a maximal use of luliconazole cream 1% to evaluate the highest systemic exposure of luliconazole, but the doses administered were higher than intended by approximately 25%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.